CLINICAL TRIAL: NCT06871085
Title: Effectiveness of a Novel Sock Design on Ankle and Postural Stability
Brief Title: Novel Sock Design on Ankle and Postural Stability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, William J. Hanney, Professor, University of Central Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00007246
Record Dates: First submitted 2025-02-13; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Ankle Stability; Postural Stability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sock (Experimental): Ankle and postural stability will be evaluated with and without use of a novel stability sock
  Interventions: Device: Stability Sock

INTERVENTIONS:
Device: Stability Sock — Use of a stability sock

SUMMARY:
This study uses a prospective cohort study design using a convenience sample to explore the sock's impact on various aspects of ankle function and overall stability. A secondary objective is measuring subjective changes in reported confidence levels in performing balance and stability exercises with and without sock

DETAILED DESCRIPTION:
Study Design: This study uses a prospective cohort design to assess the effects of wearing the novel sock on ankle stability, muscle activation, and functional performance.

Participant Consent:

All participants will provide informed consent before beginning the study. They will be given the opportunity to ask questions about the procedures and consent will be documented by both the participant and the researcher. This process will take about 5 minutes.

Participant Screening:

Each participant will undergo screening based on the inclusion/exclusion criteria. They must be 18 years or older, with no recent ankle injury or surgery and no reported feelings of ankle instability or allergies to the sock material.

A medical history questionnaire will be completed by each participant to confirm their eligibility. This process will take about 5 minutes.

Warm-up and Familiarization:

Participants will undergo the previously described warm-up, including 10 repetitions of specific exercises (toe spreads, toe raises, heel raises) and walking 120 meters to familiarize themselves with the sock. Warm-up will take 30 seconds for each exercise, and walking for familiarization will take about 1 minute.

Functional Assessments:

All assessments will be performed with and without the sock. The performance of the assessments with or without the socks will be randomized with each participant. Once randomized, all assessments will be performed and then the patient will either put on or take off the sock and perform the assessments again.

Grip Strength:

Grip strength will be measured using a hand dynamometer. Participants will sit in a chair with no armrests, feet flat on the floor, and squeeze the dynamometer with each hand while their forearm is positioned in a neutral position.

Two trials will be conducted per hand, alternating hands with a 1-minute rest between each trial. The average of the two trials will be recorded. This assessment will take about 5 minutes.

Single Leg Stance:

This test measures static balance. Participants will be asked to stand on one leg, starting with the right leg. Timing will start when the participant lifts one foot off the ground and will stop when balance is lost or the foot touches the ground again.

Each leg will be tested, and the average time from two trials will be recorded. This assessment will take about 5 minutes.

Y-Balance Test (YBT):

The YBT will be used to measure dynamic balance. Participants will stand on one leg and use the other leg to push a reach indicator in three different directions (anterior, posteromedial, and posterolateral).

Six practice trials will be done, followed by three measured trials per leg. The distances reached will be recorded, and the average of the last three trials of each leg will be taken This assessment will take about 8 minutes.

Functional Reach Standing:

Participants will stand with their arm extended at 90 degrees and reach as far forward as possible without stepping. The distance reached will be measured and recorded using a yardstick.

This test measures postural control and stability. This assessment will take about 2 minutes.

Single Leg Hop:

This test will measure dynamic balance and power. Participants will perform three types of hops: forward, lateral, and triple hops, landing on one leg. Each landing will be observed and assessed for balance. Participants will perform one practice attempt, then three trials for each test. The average of the three attempts will be recorded.

The distance for each hop and any balance errors will be recorded. This assessment will take about 8 minutes.

Balance Error Scoring System (BESS):

Participants will perform balance stances (double leg, single leg, and tandem) on both a flat surface and foam pad for 20 seconds each. The researcher will record any balance errors such as eye opening or stepping off the testing surface. This assessment will take about 3 minutes.

Fingertip to Floor Test (FFT) Participants will stand with their feet together on a 21.2 cm box and try to bend forward to reach as far down towards the floor as possible without bending their knees. Distance of fingertips from the ground will be recorded, if their fingertips touch the floor their radial styloid process will be used instead to measure the distance from the floor, using a ruler in centimeters. 1 practice trial will be conducted followed by 1 test trial. This test will take about 2 minutes to complete.

After all tests have been performed with and without the novel sock, the participants will be asked to complete a google form questionnaire about their perceptions of their performance with and without the sock.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 18 years old or older
* Able to perform the following actions with no pain or discomfort: sit-to-stand, jump, one leg stand
* Must read, write, and speak sufficient English in order to complete subjective questionnaire

Exclusion Criteria:

* Had a previous foot or leg injury
* Had a foot condition at the time of their participation in the study
* Had feelings of instability at the ankle
* Had an ankle injury within the past 12 months
* Had surgery on either lower extremity in the past
* Had any torn ligaments or cartilage at the hip, knee, or ankle
* Experienced radicular symptoms down either lower extremity
* Had any allergies to the sock material used in the study

  1. 80% nylon
  2. 14% polyester
  3. 6% elastane
* Is currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-03 (Estimated); Primary Completion 2025-08-25 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Grip Strength: | Immediately after intervention
  Grip strength will be measured using a hand dynamometer. Participants will sit in a chair with no armrests, feet flat on the floor, and squeeze the dynamometer with each hand while their forearm is positioned in a neutral position.
  Two trials will be conducted per hand, alternating hands with a 1-minute rest between each trial. The average of the two trials will be recorded. This assessment will take about 5 minutes.
Single Leg Stance | Immediately after intervention
  This test measures static balance. Participants will be asked to stand on one leg, starting with the right leg. Timing will start when the participant lifts one foot off the ground and will stop when balance is lost or the foot touches the ground again.
  Each leg will be tested, and the average time from two trials will be recorded. This assessment will take about 5 minutes.
Y-Balance Test (YBT) | Immediately after intervention
  The YBT will be used to measure dynamic balance. Participants will stand on one leg and use the other leg to push a reach indicator in three different directions (anterior, posteromedial, and posterolateral).
  Six practice trials will be done, followed by three measured trials per leg. The distances reached will be recorded, and the average of the last three trials of each leg will be taken This assessment will take about 8 minutes.
Functional Reach Standing | Immediately after intervention
  Participants will stand with their arm extended at 90 degrees and reach as far forward as possible without stepping. The distance reached will be measured and recorded using a yardstick.
  This test measures postural control and stability. This assessment will take about 2 minutes.
Single Leg Hop | Immediately after intervention
  This test will measure dynamic balance and power. Participants will perform three types of hops: forward, lateral, and triple hops, landing on one leg. Each landing will be observed and assessed for balance. Participants will perform one practice attempt, then three trials for each test. The average of the three attempts will be recorded.
  The distance for each hop and any balance errors will be recorded. This assessment will take about 8 minutes.
Balance Error Scoring System (BESS) | Immediately after intervention
  Participants will perform balance stances (double leg, single leg, and tandem) on both a flat surface and foam pad for 20 seconds each. The researcher will record any balance errors such as eye opening or stepping off the testing surface. This assessment will take about 3 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upon request

REFERENCES:
- [Background] Taylor JB, Wright ES, Waxman JP, Schmitz RJ, Groves JD, Shultz SJ. Ankle Dorsiflexion Affects Hip and Knee Biomechanics During Landing. Sports Health. 2022 May-Jun;14(3):328-335. doi: 10.1177/19417381211019683. Epub 2021 Jun 6. PMID 34096370